CLINICAL TRIAL: NCT05094791
Title: Lateralization After IntraMedullary Nailing of InterTrochanteric Hip Fractures, Clinical and Radiographic Outcomes
Acronym: LIMIT
Status: Completed | Type: Observational
Sponsor: Prisma Health-Upstate (Other)
Collaborators: Arthrex, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00113048
Record Dates: First submitted 2021-10-04; First posted 2021-10-26 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Intertrochanteric Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- Telescoping Lag Screw: Intertrochanteric fractures treated with Arthrex Hip Nail with Telescoping Screw
  Interventions: Device: Telescoping Lag Screw
- Standard lag Screw: Intertrochanteric fractures treated with Zimmer Natural Nail Cephalomedullary Nail
  Interventions: Device: Standard lag Screw
- Standard lag screw with addition of worm screw: Intertrochanteric fractures treated with Smith and Nephew TRIGEN INTERTAN
  Interventions: Device: Standard lag screw with addition of worm screw

INTERVENTIONS:
Device: Telescoping Lag Screw — Intertrochanteric fracture fixation using Arthrex Hip Nail with Telescoping Lag Screw
  Other Names: Arthrex Hip Nail
  Groups: Telescoping Lag Screw
Device: Standard lag Screw — Intertrochanteric fracture fixation using Zimmer Natural Nail Cephalomedullary Nail using standard lag screw
  Other Names: Zimmer Natural Nail
  Groups: Standard lag Screw
Device: Standard lag screw with addition of worm screw — Intertrochanteric fracture fixation using Smith and Nephew TRIGEN INTERTAN with addition of worm screw
  Other Names: Smith and Nephew TRIGEN INTERTAN
  Groups: Standard lag screw with addition of worm screw

SUMMARY:
Intertrochanteric fractures are commonly stabilized using an intramedullary nail with a lag screw that enters the lateral cortex of the femur. This lag screw commonly protrudes during the healing process and may cause implant related pain. This study will help determine if implant related pain is different depending to the lag screw design.

DETAILED DESCRIPTION:
This study compares cephalomedullary fixation of intertrochanteric femur fractures using the Arthrex Hip Nail System with a telescoping lag screw compared to the Zimmer Natural Nail and the Smith and Nephew InterTan. This pilot study will evaluate radiographic outcomes and lateral sided hip pain related to different lag screw designs used for patients with intertrochanteric femur fractures by comparing outcomes of patients receiving 3 different lag screws The primary objective of this study is to compare pain at the level of the lag screw of patients with collapsible lag screws compared to patient who received a standard lag screw using a numeric rating scale on a 0-100 scale.

ELIGIBILITY:
Inclusion Criteria:

* Patients greater than or equal to 22 years of age who undergo treatment of an intertrochanteric hip fracture with an intramedullary nail.
* Fluoroscopic views of the final fixation construct or a post-operative radiograph taken within 24 hours must be available.

Exclusion Criteria:

* Non-ambulatory prior to injury (patient must do more than only transfers)
* Cognitive deficiencies that prevent the patient from providing their own informed consent
* Inability to follow-up at the discretion of the investigator (incarceration, moving out of area, no permanent housing)
* Prior fracture to injured hip
* Prior surgery to injured hip
* Basi-cervical fracture pattern (fracture that begins above the lesser trochanter and exits medial to the greater trochanter)
* Patients not treated within 48 hours of admission
* Chronic or acute infection at site of surgery
* Language barrier preventing completion of study forms in English
* Open fracture
* Fracture related to neoplasm

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients sustaining an intertrochantic hip fracture
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-02-23 (Actual)

PRIMARY OUTCOMES:
Pain at lag screw | 6 weeks
  Pain will be accessed at the location of the lag screw, pain will be measured by using a Numeric rating scale (0-100)
Pain at lag screw | 12 weeks
  Pain will be accessed at the location of the lag screw, pain will be measured by using a Numeric rating scale (0-100)
Pain at lag screw | 21 weeks
  Pain will be accessed at the location of the lag screw, pain will be measured by using a Numeric rating scale (0-100)
Pain at lag screw | 52 weeks
  Pain will be accessed at the location of the lag screw, pain will be measured by using a Numeric rating scale (0-100)

SECONDARY OUTCOMES:
Radiographic lateralization of lag screw | 52 weeks
  Change in the lateralization of the lag screw measured in mm
Incidence of lag screw injections | 52 weeks
  Incidence of patients requiring injections at the location of the lag screw due to pain
Reoperation rate | 52 weeks
  Reoperations to the location in the intertrochanteric fractue

CONTACTS AND LOCATIONS:
Overall Officials: John D Adams, MD, Principal Investigator — Prisma Health
Locations (1):
- Greenville Memorial Hosptial, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No